CLINICAL TRIAL: NCT05376748
Title: Exercise Capacity in Patients With Heart Failure With Preserved Ejection Fraction Before and After Ablation of Atrial Fibrillation
Brief Title: Exercise Capacity Before and After AF Ablation in Patients With HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Nicole Habel, MD, Principal Investigator, University of Vermont
Other Study IDs: 00001607
Record Dates: First submitted 2022-04-25; First posted 2022-05-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Atrial Fibrillation
Keywords: Ablation; HFpEF; atrial fibrillation; exercise capacity; peak oxygen consumption
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
In a prospective, observational pilot study of patients scheduled for an atrial fibrillation (AF) ablation at the University of Vermont Medical Center the investigators will compare exercise capacity before and four months after AF ablation.

DETAILED DESCRIPTION:
Patients ≥ 18 years of age who are scheduled for an AF ablation at the University of Vermont Medical Center will be screened for the following inclusion criteria: H2FpEF score of ≥ 6 (corresponding to ≥90% probability of HFpEF (19)) AND echocardiogram within the past 2 years that reported a LV ejection fraction ≥ 50% AND at least one symptom of HF (dyspnea on exertion, orthopnea or paroxysmal nocturnal dyspnea). Exclusion criteria: (1) Life expectancy <12 months, (2) moderate or more valvular disease, (3) inability to walk on a treadmill. Patients with early recurrent AF (defined as AF after a 12-week post-procedural blanking period accounting for post-ablation inflammation) will be withdrawn from the study and not proceed to the 4 month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* H2FpEF score of ≥ 6 (corresponding to >90% probability of HFpEF (19))
* echocardiogram within the past 2 years that reported a LV ejection fraction ≥ 50%
* at least one symptom of HF (dyspnea on exertion, orthopnea or paroxysmal nocturnal dyspnea).
* AF ablation scheduled at UVMMC

Exclusion Criteria:

* Life expectancy <12 months
* moderate or more valvular disease
* inability to walk on a treadmill

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with atrial fibrillation and HFpEF who are undergoing AF ablation
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in peak VO2 | before AF ablation and 4 months after AF ablation
  cardiopulmonary exercise testing will be performed & peak VO2 measured at baseline & follow up visit

SECONDARY OUTCOMES:
Change in KCCQ score | before and 4 months after AF ablation
  Kansas City Cardiomyopathy Questionnaire (KCCQ) will be obtained at baseline visit & again at ablation follow up visit. Scale 0-100 with higher scores signifying better quality of life.
Percent change in NTproBNP | before and 4 months after AF ablation
  Initial sample taken day of AF ablation as is standard of care; reassessed at 4 month f/u visit

OTHER OUTCOMES:
Difference in peak VO2 in patient with vs. without chronic rate control | 4 months post-ablation
  4 months f/u cardiopulmonary exercise testing performance compared between those with and without chronic rate control

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Habel, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oktay AA, Rich JD, Shah SJ. The emerging epidemic of heart failure with preserved ejection fraction. Curr Heart Fail Rep. 2013 Dec;10(4):401-10. doi: 10.1007/s11897-013-0155-7. PMID 24078336
- [Background] Vasan RS, Benjamin EJ, Levy D. Prevalence, clinical features and prognosis of diastolic heart failure: an epidemiologic perspective. J Am Coll Cardiol. 1995 Dec;26(7):1565-74. doi: 10.1016/0735-1097(95)00381-9. PMID 7594087
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Haykowsky MJ, Brubaker PH, John JM, Stewart KP, Morgan TM, Kitzman DW. Determinants of exercise intolerance in elderly heart failure patients with preserved ejection fraction. J Am Coll Cardiol. 2011 Jul 12;58(3):265-74. doi: 10.1016/j.jacc.2011.02.055. PMID 21737017
- [Background] Mikkelsen N, Cadarso-Suarez C, Lado-Baleato O, Diaz-Louzao C, Gil CP, Reeh J, Rasmusen H, Prescott E. Improvement in VO2peak predicts readmissions for cardiovascular disease and mortality in patients undergoing cardiac rehabilitation. Eur J Prev Cardiol. 2020 May;27(8):811-819. doi: 10.1177/2047487319887835. Epub 2019 Nov 19. PMID 31744334
- [Background] Swank AM, Horton J, Fleg JL, Fonarow GC, Keteyian S, Goldberg L, Wolfel G, Handberg EM, Bensimhon D, Illiou MC, Vest M, Ewald G, Blackburn G, Leifer E, Cooper L, Kraus WE; HF-ACTION Investigators. Modest increase in peak VO2 is related to better clinical outcomes in chronic heart failure patients: results from heart failure and a controlled trial to investigate outcomes of exercise training. Circ Heart Fail. 2012 Sep 1;5(5):579-85. doi: 10.1161/CIRCHEARTFAILURE.111.965186. Epub 2012 Jul 6. PMID 22773109
- [Background] Nadruz W Jr, West E, Sengelov M, Santos M, Groarke JD, Forman DE, Claggett B, Skali H, Shah AM. Prognostic Value of Cardiopulmonary Exercise Testing in Heart Failure With Reduced, Midrange, and Preserved Ejection Fraction. J Am Heart Assoc. 2017 Oct 31;6(11):e006000. doi: 10.1161/JAHA.117.006000. PMID 29089342
- [Background] Reddy YNV, Obokata M, Verbrugge FH, Lin G, Borlaug BA. Atrial Dysfunction in Patients With Heart Failure With Preserved Ejection Fraction and Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1051-1064. doi: 10.1016/j.jacc.2020.07.009. PMID 32854840
- [Background] Elshazly MB, Senn T, Wu Y, Lindsay B, Saliba W, Wazni O, Cho L. Impact of Atrial Fibrillation on Exercise Capacity and Mortality in Heart Failure With Preserved Ejection Fraction: Insights From Cardiopulmonary Stress Testing. J Am Heart Assoc. 2017 Oct 31;6(11):e006662. doi: 10.1161/JAHA.117.006662. PMID 29089343
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Belardinelli R, Georgiou D, Cianci G, Purcaro A. Randomized, controlled trial of long-term moderate exercise training in chronic heart failure: effects on functional capacity, quality of life, and clinical outcome. Circulation. 1999 Mar 9;99(9):1173-82. doi: 10.1161/01.cir.99.9.1173. PMID 10069785
- [Background] Tamargo M, Obokata M, Reddy YNV, Pislaru SV, Lin G, Egbe AC, Nishimura RA, Borlaug BA. Functional mitral regurgitation and left atrial myopathy in heart failure with preserved ejection fraction. Eur J Heart Fail. 2020 Mar;22(3):489-498. doi: 10.1002/ejhf.1699. Epub 2020 Jan 7. PMID 31908127
- [Background] Kaye DM, Silvestry FE, Gustafsson F, Cleland JG, van Veldhuisen DJ, Ponikowski P, Komtebedde J, Nanayakkara S, Burkhoff D, Shah SJ. Impact of atrial fibrillation on rest and exercise haemodynamics in heart failure with mid-range and preserved ejection fraction. Eur J Heart Fail. 2017 Dec;19(12):1690-1697. doi: 10.1002/ejhf.930. Epub 2017 Oct 11. PMID 29024227
- [Background] Fukasawa K, Fukuda K, Mori N, Kondo M, Chiba T, Miki K, Hasebe Y, Nakano M, Shimokawa H. Impacts of sinus rhythm maintenance with catheter ablation on exercise tolerance in patients with paroxysmal atrial fibrillation. J Interv Card Electrophysiol. 2021 Jun;61(1):105-113. doi: 10.1007/s10840-020-00786-y. Epub 2020 Jun 1. PMID 32488748
- [Background] Di Biase L, Mohanty P, Mohanty S, Santangeli P, Trivedi C, Lakkireddy D, Reddy M, Jais P, Themistoclakis S, Dello Russo A, Casella M, Pelargonio G, Narducci ML, Schweikert R, Neuzil P, Sanchez J, Horton R, Beheiry S, Hongo R, Hao S, Rossillo A, Forleo G, Tondo C, Burkhardt JD, Haissaguerre M, Natale A. Ablation Versus Amiodarone for Treatment of Persistent Atrial Fibrillation in Patients With Congestive Heart Failure and an Implanted Device: Results From the AATAC Multicenter Randomized Trial. Circulation. 2016 Apr 26;133(17):1637-44. doi: 10.1161/CIRCULATIONAHA.115.019406. Epub 2016 Mar 30. PMID 27029350
- [Background] Marrouche NF, Brachmann J, Andresen D, Siebels J, Boersma L, Jordaens L, Merkely B, Pokushalov E, Sanders P, Proff J, Schunkert H, Christ H, Vogt J, Bansch D; CASTLE-AF Investigators. Catheter Ablation for Atrial Fibrillation with Heart Failure. N Engl J Med. 2018 Feb 1;378(5):417-427. doi: 10.1056/NEJMoa1707855. PMID 29385358
- [Background] Reddy YNV, Carter RE, Obokata M, Redfield MM, Borlaug BA. A Simple, Evidence-Based Approach to Help Guide Diagnosis of Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):861-870. doi: 10.1161/CIRCULATIONAHA.118.034646. PMID 29792299
- [Background] Kitzman DW, Brubaker PH, Morgan TM, Stewart KP, Little WC. Exercise training in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. Circ Heart Fail. 2010 Nov;3(6):659-67. doi: 10.1161/CIRCHEARTFAILURE.110.958785. Epub 2010 Sep 17. PMID 20852060
- [Background] Sugumar H, Nanayakkara S, Vizi D, Chieng D, Leet A, Mariani J, Taylor A, Kalman J, Kistler P, Ling L. Impact of catheter ablation on HFpEF in people with comorbid atrial fibrillation and HFpEF using invasive haemodynamic testing. European Heart Journal. 2020; 41(2): ehaa946.0892.